CLINICAL TRIAL: NCT01289353
Title: Phase I-II Study of Concurrent Adjuvant Systemic Therapy and Accelerated Radiotherapy (Over 3 Weeks)
Brief Title: Concurrent Adjuvant Carboplatin and Accelerated Radiotherapy for Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-01969
Record Dates: First submitted 2011-01-31; First posted 2011-02-03 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
Keywords: triple negative; breast cancer; adjuvant therapy; Carboplatin; chemotherapy; radiation therapy; chemo-radiotherapy; accelerated radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ChemoRT (Experimental): Concurrent Carboplatin and Radiotherapy
  Interventions: Drug: Carboplatin; Radiation: 3D-RT or IMRT

INTERVENTIONS:
Drug: Carboplatin — IV, weekly for 6 weeks, AUC of 2.0
  Other Names: Paraplatin
Radiation: 3D-RT or IMRT — From week 2 to week 4 in the 6-week Carboplatin treatment:
  Whole Breast 3D-RT or IMRT at 2.7 Gy X 15 fractions (5 times/wk x 3 wks=40.50 Gy), then the second and third Friday, 3 Gy to the tumor bed only X 2 fractions, Total dose to tumor bed = 46.5 Gy

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of a combination of chemotherapy and radiotherapy in breast cancer patients after breast surgery.

DETAILED DESCRIPTION:
Preliminary experience in the neo-adjuvant setting of Locally Advanced Breast Cancer (LABC) has recently demonstrated that hormone receptors negative patients have approximately 50% chance to achieve a pathological response after concurrent chemo-radiation. In a multi-institutional collaboration of 105 patients it was found that triple negative (TN) tumor carriers achieved pathological response in 54% of the cases and that the response reflected on 5-year disease free survival and overall survival. Our group has speculated that these effects on the risk of distant recurrence could depend on the recovery of antitumor immunity among the patients achieving pathological response, after tumor cell death induced by concurrent chemo-radiation.

The investigators are proposing a novel study that translates these findings to the adjuvant setting of TN tumors. TN breast cancer is a more aggressive form of the disease often coinciding with basal-like tumors. BRCA mutated-cancer is more frequently TN.

The current protocol converges the experience NYU has developed in accelerated prone breast radiotherapy with encouraging finding from the use of concurrent chemoradiation in LABC.

The investigators will study the feasibility of combining weekly carboplatin with concurrent 3-weeks prone breast radiotherapy in the adjuvant setting of 35 women with TN tumors, after segmental mastectomy and nodal assessment. Primary endpoint of the study is acute toxicity of the combined regimen, with a target of < 25% of grade II-III dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18
* Pre- or post-menopausal women with Stage I and II breast cancer, triple negative tumors
* Biopsy-proven invasive breast cancer, excised with negative margins of at least 1 mm
* Status post segmental mastectomy, after sentinel node biopsy and/or axillary node dissection (Tumors < 5 mm in size do not require nodal assessment) or after mastectomy
* No previous chemotherapy
* Patient needs to be able to understand and demonstrate willingness to sign a written informed consent document

Exclusion Criteria:

* Previous radiation therapy to the ipsilateral breast
* Active connective tissue disorders, such as lupus or scleroderma
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-03-06 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Perez, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ChemoRT
Started | 92
Completed | 90
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | ChemoRT
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.83 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 20
  More than one race | 0
  Unknown or Not Reported | 57
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Developed Grade 2-3 Acute Radiation Dermatitis Within 60 Days Post-RT
Time Frame: 60 days post-RT
Measure: Count of Participants; unit: Participants
Arm/Group | ChemoRT
Number analyzed (Participants) | 90
Participants | 8

2. Secondary Outcome: Number of Patients Who Experience Acute Toxicities at or More Than 6 Months After Completion of Radiation Treatment (RT)
Description: Acute Toxicities include all Grade 1 toxicities
Time Frame: 6 months to 5 year post-RT
Measure: Count of Participants; unit: Participants
Arm/Group | ChemoRT
Number analyzed (Participants) | 90
Participants | 67

3. Secondary Outcome: Number of Patients Who Experience Grade 2 or Higher Late Toxicities at or More Than 6 Months After Completion of Radiation Treatment (RT)
Time Frame: 6 months to 5 years post-RT
Measure: Count of Participants; unit: Participants
Arm/Group | ChemoRT
Number analyzed (Participants) | 90
Participants | 18

ADVERSE EVENTS:
Time Frame: 5 years post-RT
Arm/Group | ChemoRT
All-Cause Mortality (participants affected / at risk) | 6/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT01289353/Prot_SAP_000.pdf